CLINICAL TRIAL: NCT04061200
Title: Renal Effects of Treatment With Empagliflozin Alone or in Combination With Semaglutide in Patients With Type 2 Diabetes and Albuminuria - A Double Blinded, Randomised, Placebo Controlled, Parallel, Single Center Study
Brief Title: Renal Effects of Treatment With Empagliflozin Alone or in Combination With Semaglutide in Patients With Type 2 Diabetes and Albuminuria
Acronym: EmpaSema
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-003175-19
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes With Renal Manifestations
MeSH Terms: interventions — semaglutide; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide 1,34 mg/ml (Active Comparator): Semaglutide 1,34 mg/ml (solution for subcutaneous injection in pre-filled pen-injector). At randomisation, the participants start with doses of 0.25 mg/week for 4 weeks, then escalate to doses of 0.5 mg/week for 4 weeks, and thereafter escalate to 1.0 mg/week if tolerated until 52 weeks of total treatment.
  Interventions: Drug: Semaglutide, 1.34 mg/mL; Other: Placebo, 1,34 mg/mL; Drug: Empagliflozin 25 MG
- Placebo 1,34 mg/ml (Placebo Comparator): Placebo 1,34 mg/ml (solution for subcutaneous injection in pre-filled pen-injector). At randomisation, the participants start with doses of 0.25 mg/week for 4 weeks, then escalate to doses of 0.5 mg/week for 4 weeks, and thereafter escalate to 1.0 mg/week if tolerated until 52 weeks of total treatment.
  Interventions: Drug: Semaglutide, 1.34 mg/mL; Other: Placebo, 1,34 mg/mL; Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Semaglutide, 1.34 mg/mL — After informed consent, subjects will be initiated on open-label empagliflozin 25 mg or maximal tolerated dosis once daily during a run-in period of 26 weeks. Participants will be randomized and up titrated to semaglutide 1.34 mg/ml or matching placebo once weekly during the following 26 weeks in a 1:1 ratio.
Other: Placebo, 1,34 mg/mL — Participants will be randomised to either semaglutide or placebo as an add on treatment after 26 weeks of intervention with empagliflozin 25 mg.
Drug: Empagliflozin 25 MG — After informed consent, subjects will be initiated on open-label empagliflozin 25 mg or maximal tolerated dosis once daily during a run-in period of 26 weeks.

SUMMARY:
The objective of this study is to evaluate the effect of treatment with semaglutide 1.34 mg/ml in combination with empagliflozin 25 mg, compared to treatment with empagliflozin 25 mg in combination with placebo on albuminuria in participants with type 2 diabetes and albuminuria.

In a randomised, placebo-controlled, double-blinded, parallel trial we will include 80 patients with type 2 diabetes and albuminuria. Patients will start in a run-in phase of 26 weeks with empagliflozin 25 mg alone. After that, the patients will be randomised 1:1 to an active treatment period with semaglutide of 26 weeks or placebo for 26 weeks.

The primary endpoint is change from randomisation to week 52 in albuminuria, measured in three morning urine samples.

DETAILED DESCRIPTION:
Patients with type 2 diabetes are at high risk of developing diabetic nephropathy. The most promising antidiabetic agents on the market with potential to preserve renal function are endogenous glucagon like peptide (GLP-1) agonists and selective sodium-glucose cotransporter 2 (SGLT2) inhibitors. The LEADER trial demonstrated that treatment with liraglutide (GLP-1 agonist) resulted in 22% lower risk of renal composite outcome. The EMPA-REG trial demonstrated that treatment with empagliflozin (SGLT2 inhibitor) reduced the same renal composite outcome by 39%.

Previous studies have mainly focused on glycaemic parameters when combining a GLP-1 agonist and SGLT2 inhibitor. From a renal perspective, it is of major interest to investigate if a stepwise initiation of semaglutide or placebo added to ongoing empagliflozin therapy would complement or have an additive effect on renal parameters.

In a randomised, placebo-controlled, double-blinded, parallel trial we will include 80 patients with type 2 diabetes and albuminuria. Patients will start in a run-in phase of 26 weeks with empagliflozin 25 mg alone. After that, the patients will be randomised 1:1 to an active treatment period with semaglutide of 26 weeks or placebo for 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Given written informed consent
2. Male or female patients ≥ 18 years with type 2 diabetes (WHO criteria).
3. UACR > 100 mg/g within a year of informed consent documented in the medical files.
4. eGFR ≥ 30 ml/min/1.73 m2 (estimated by CKD-EPI formula) within 3 months of informed consent documented in the medical files. The eGFR measured at visit 0 has to meet the criteria as well.
5. Fertile female must use chemical, hormonal and mechanical contraceptives, be in menopause (i.e. must not have had regular menstrual bleeding for at least one year), have undergone bilateral oophorectomy or have been surgically sterilized or hysterectomised at least six months prior to screening
6. Treated with maximal tolerated dose of an angiotensin-converting-enzyme inhibitor or an angiotensin II receptor blocker, 4 weeks prior to randomisation. If the participants are not treated with maximal tolerated dosis the investigator will increase the dose 4 weeks prior randomisation if tolerated.
7. Ability to communicate with the investigator and understand informed consent.

Exclusion Criteria:

1. Type 1 diabetes
2. Known or suspected hypersensitivity to trial product(s) or related products
3. Cancer (except basal cell skin cancer or squamous cell skin cancer) or any other clinically significant disorder, except for conditions associated with type 2 diabetes history, which in the investigators opinion could interfere with the results of the trial
4. Cardiac disease defined as: Decompensated heart failure (NYHA class III-IV) and or diagnosis of unstable angina pectoris and/or myocardial infarction within the last 6 months.
5. Previous bowel resection
6. Body mass index < 18.5 kg/m2
7. Females of childbearing potential who are pregnant, breast-feeding, intend to become pregnant or are not using adequate contraceptive methods
8. Known or suspected abuse of alcohol or narcotics.
9. Participant in another intervention study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Albuminuria | From randomisation to week 52
  Change in albuminuria

SECONDARY OUTCOMES:
Hba1c | From randomisation to week 52
  Change in Hba1c
GFR | From randomisation to week 52
  Change in measured kidney function (GFR)
24 hour blood pressure | From randomisation to week 52
  Change in 24 hour blood pressure
Vasoactive hormones | From randomisation to week 52
  Change in vasoactive hormones (o Plasma renin concentration, plasma renin activity, angiotensin I, angiotensin II, aldosterone, copeptin)
Inflammatory and endothelial biomarkers | From randomisation to week 52
  Change in inflammatory and endothelial biomarkers (Von Willebrand factor, sVCAM-1, sICAM-1, E-selectin, b-leucocytes, s-CRP, IL-6, osteopontin, TNF-α)

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818